CLINICAL TRIAL: NCT05851885
Title: A Single-center, Prospective, Parallel Randomized Controlled Study Evaluating the Clinical Effectiveness of an Intelligent Graphic Report System for Upper Gastrointestinal Endoscopy
Brief Title: Evaluation of the Clinical Effectiveness of Upper Gastrointestinal Endoscopy Reporting System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EA-23-007
Record Dates: First submitted 2023-04-30; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Endoscopy, Gastrointestinal; Artificial Intelligence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Physicians draft EGD reports with the assistance of the AI-based reporting system.
  Interventions: Diagnostic Test: AI-based reporting system
- Control group (No Intervention): Physicians use the conventional reporting system to draft EGD reports. At the same time, the AI-based reporting system will automatically generate a report of the EGD examination.

INTERVENTIONS:
Diagnostic Test: AI-based reporting system — AI-based reporting system is a software platform for real-time analysis and records of abnormalities and landmarks during endoscopy.
  Arms: Experimental group

SUMMARY:
The objective of this study is to assess the effectiveness of an AI-based reporting system for upper gastrointestinal endoscopy. The primary question that this study aims to address is whether the reporting system can enhance the completeness and accuracy of endoscopic reports when assisted by AI, as drafted by endoscopists. Patients will be randomly assigned to either the experimental group or the control group. In the experimental group, physicians will draft EGD reports with the assistance of the AI-based reporting system, while in the control group, physicians will use the conventional reporting system to draft EGD reports. At the same time, the AI-based reporting system will automatically generate a report of the EGD examination.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years
2. Aim to undergo screening, surveillance, and diagnosis
3. Undergo sedated EGD
4. Able to read, understand, and sign informed consent

Exclusion Criteria:

1. EGD contraindications
2. Not suitable for sedated endoscopy after anaesthesia evaluation
3. Biopsy contraindications
4. Active upper gastrointestinal bleeding or emergency oesophagogastroduodenoscopy (EGD)
5. Pregnancy
6. Upper gastrointestinal surgery or residual stomach
7. Not suitable for recruitment after investigator evaluation because of other high-risk conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Completeness of reporting lesions | one month
  Calculation method = number of report lesions / total number of lesions x 100%

SECONDARY OUTCOMES:
Completeness of report drafting on lesion features | one month
  Calculation method = number of drafted features of lesions / total number of features required to be drafted x 100%
Accuracy of report drafting on lesion features | one month
  Calculation method = number of accurately drafted features of lesions / total number of drafted features x 100%
Reporting time | one month
  The time that endoscopists draft reports
Completeness of reporting lesions of AI system | one month
  Calculation method = number of report lesions / total number of lesions x 100%
Accuracy of report drafting on lesion features of AI system | one month
  Calculation method = number of accurately drafted features of lesions / total number of drafted features x 100%
Physician satisfaction survey | one month
  Use 5-point Likert scale to assess physician satisfaction, acceptance, and trust in using the intelligent graphic report system to draft endoscopic reports.

CONTACTS AND LOCATIONS:
Overall Officials: Honggang Yu, MD, Principal Investigator — Wuhan University Renmin Hospital